CLINICAL TRIAL: NCT01981694
Title: A Phase 1, Double Blind, Sponsor Open, Randomized, Placebo Controlled, Crossover, Single Oral Dose Escalation Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of PF-06649751 in Healthy Subjects
Brief Title: A Phase I Trial to Investigate the Safety and Tolerability of PF-06649751
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B7601001
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: Phase 1; Randomized; Double Blind; Placebo-Controlled; Single-Dose Escalation; Safety; Tolerability; PK; PD; PF-06649751

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single ascending doses (Experimental)
  Interventions: Drug: PF-06649751
- Measurement of eye blink rate (Experimental)
  Interventions: Drug: PF-06649751

INTERVENTIONS:
Drug: PF-06649751 — Single doses, given by oral solution, starting at 0.25 mg up to a possible maximum of 7.5 mg. The subject will have been fasted for 10 hours prior to the single dose. For each dosing period, 3 subjects will be given a placebo as a comparator. One dose will be given in the fed state.
  Arms: Single ascending doses
Drug: PF-06649751 — It is believed that the maximum tolerated dose of this compound the eye blink rate (EBR) will also increase. This arm will use EBR measurement technology to verify this hypothesis. In each dosing period, 5 subjects will be given a placebo as a comparator.
  Arms: Measurement of eye blink rate

SUMMARY:
This study will determine the safety and tolerability of PF-06649751 given orally to healthy volunteers. To determine the optimal dose for future studies, the concentration of the drug over time will be determined by periodic blood samples. The rate of eye blinks will be measured as an indicator of PF-06649751 action on the receptors of interest in the brain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non-childbearing potential between the ages of 18 and 55 years
* Female subjects of non childbearing potential that meet at least one of the following criteria: Achieved postmenopausal status, defined as: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and have a serum follicle stimulating hormone (FSH) level confirming the postmenopausal status; Have undergone a documented hysterectomy and/or bilateral oophorectomy; Have medically confirmed ovarian failure.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption.
* Subjects with epilepsy, or history of epilepsy, or conditions that lower seizure threshold, seizures of any etiology (including substance or drug withdrawal), or who have increased risk of seizures as evidenced by history of EEG with epileptiform activity. Subjects with a history of childhood seizures, and history of head trauma with loss of consciousness requiring hospitalization overnight will be excluded as well.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 16, 24, 32, 48, 72 hours post-dose
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 0, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 16, 24, 32, 48, 72 hours post-dose
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Maximum Observed Plasma Concentration (Cmax) | 0, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 16, 24, 32, 48, 72 hours post-dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 16, 24, 32, 48, 72 hours post-dose
Plasma Decay Half-Life (t1/2) | 0, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 16, 24, 32, 48, 72 hours post-dose
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Apparent Oral Clearance (CL/F) | 0, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 16, 24, 32, 48, 72 hours post-dose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) | 0, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 16, 24, 32, 48, 72 hours post-dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Eye Blink Rate | 0, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 16, 24 hours post-dose
  Measurement of eye blink rate for a given dose at time of predicted maximum blood concentration of the compound

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7601001&StudyName=A%20Phase%20I%20Trial%20to%20Investigate%20the%20Safety%20and%20Tolerability%20of%20PF-06649751